CLINICAL TRIAL: NCT04001686
Title: Ambispective Observational Study to Evaluate the Incidence and Management of Aplastic Anemia in Spain
Acronym: IISAPM201701
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Biogipuzkoa Health Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: IIS-APM-2017-01
Record Dates: First submitted 2019-06-26; First posted 2019-06-28 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-07

CONDITIONS: Aplastic Anemia
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: incidence aplastic anemia — Ambispective chart review

SUMMARY:
This is a national, multicenter, ambispective, observational post-authorization study (EPA-SP for its acronym in Spanish) to describe the incidence, clinical management and outcome of aplastic anemia in hospitals throughout Spain.

DETAILED DESCRIPTION:
This is a national, multicenter, ambispective, observational post-authorization study (EPA-SP for its acronym in Spanish) to describe the incidence, clinical management and outcome of aplastic anemia in hospitals throughout Spain.

The study includes a retrospective chart review to identify all cases of aplastic anemia diagnosed between January 2010 and the date of the study initiation and a prospective study to detect new cases of aplastic anemia during an 18-month period since the study initiation in the participant hospitals. The study is also designed to collect both retrospective and prospective data on clinical management and outcome of patients with confirmed aplastic anemia. All patients included in the study, including those cases of aplastic anemia identified since 2010 until the study initiation through the retrospective chart review that are alive at the time of inclusion in the study, will be followed up until death or lost-to-follow-up or until 6 months after the last patient is enrolled in the study.

The study consists of a baseline visit, follow-up visits every 6 months (± 15 days) until death or lost-to follow-up or up to 6 months after the last patient is enrolled in the study, and a final visit (final/premature withdrawal visit) which will be performed at the study end (6 months after the last patient is enrolled) or in case of premature withdrawal, except for patient withdrawal of consent, loss-to-follow-up or death.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes and of any age
* Confirmed diagnosis of spinal cord aplasia, regardless of its severity (moderate, severe or very serious), from January 1, 2010 (until the beginning of the study) (retrospective study) and during the inclusion period of 18 months in hospitals Participants (prospective study).

Aplasia is defined by a cellularity of the bone marrow <25% and the presence of less than the following: (i) hemoglobin <100 g / l (ii) platelet count <50 x109 / l (iii) Neutrophil count < 1.5 x 109 / l.

* Any severity of the disease according to hematological and spinal criteria (5): moderate aplasia (absolute neutrophil count [ANC]> 0.5 x 109 / l), severe (ANC 0.2-≤0.5) x 109 / l) or very severe (RAN <0.2 x 109 / l).
* Patients who voluntarily understand and sign the informed consent (if it can be provided), preferably in writing or orally before a witness, or will be obtained from the legal representative of the patient (for children under 16 years of age) before the start of the study. The deceased patients and the patients with whom they can not be contacted or have lost their follow-up, who have been diagnosed since January 1, 2010 until the beginning of the study, are exempt from the requirement of consent.

Exclusion Criteria:

* Patients with any medical or psychological alteration that, in the opinion of the investigator, could compromise the patient's ability to grant their informed consent.
* Evidence of Fanconi anemia, dyskeratosis congenita, congenital spinal cord syndrome, and myelodysplastic syndrome.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of all consecutive patients diagnosed with aplastic anemia between January 2010 and the date of finalization of the 18-month inclusion period
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the incidence of aplastic anemia | 2010-2022
  The primary endpoint of the study is the number of cases of aplastic anemia per year recorded in the databases of the participant hospitals from January 2010 and the date of the study initiation (retrospective analysis) and all new cases of aplastic anemia detected per year (prospective analysis) during an 18-month period since study initation.

SECONDARY OUTCOMES:
1. Number of patients diagnosed with moderate and severe aplastic anemia. | 2010-2022
  o The number of patients diagnosed with moderate and severe aplastic anemia will calculated. The number of cases per one million people per year will be presented.
2. Number of patients diagnosed with aplastic anemia according to their age and sex. | 2010-2022
  The number of males and females diagnosed with aplastic anemia per one million people per year will be calculated.
  The number of patients diagnosed with aplastic anemia in each age category considered (in the statistical plan) per one million people per year will be calculated.
3. Type of treatment prescribed as first-line, second-line or further-line treatment for aplastic anemia | 2010-2022
  The percentage of patients receiving each type of treatment for aplastic anemia (stem cell transplantation, immunosuppressive treatment [ATG + CSA, CSA alone], androgens, eltrombopag, etc.) for first-line, second and further lines of treatment will be calculated
4. Percentage of responder patients 90, 180, 270 and 360 days after each treatment initiation. | 2010-2022
  Hematological response will be assessed on the basis of hemoglobin, platelet and absolute neutrophil count every 3 months (90 days) according to routine clinical practice.
  Hematological response will be classified as response (CR and PR vs. NR). CR and PR to treatment will be defined as follows:
  CR: haemoglobin levels ≥120 g/L, platelet count ≥100 x 109/L, and neutrophil count ≥1.5 x 109/L.
  PR: haemoglobin levels ≥80 g/L, platelet count ≥20 x 109/L (transfusion independent), and neutrophil count ≥0.5 x 109/L.
5. Best hematological response during each treatment line (CR, PR, and NR). | 2010-2022
  Percentage of patients with CR, PR and NR as the best hematological response during each treatment line and the 95% CI will be calculated.
6. Overall survival, defined as the time elapsed since first-line treatment initiation until death from any cause. | 2010-2022
  The OS will be calculated as the time elapsed from first-line treatment initiation to death. Patients will be censored at the date of last follow-up if still alive at the time of the analysis. The probability of OS will be estimated using the Kaplan-Meier method. Median OS (range) and 95% CI will be calculated.
7. Relapse-free survival, defined as the time elapsed since complete or partial remission achievement until relapse or death from any cause | 2010-2022
  RFS will be calculated as the time elapsed since complete or partial remission achievement until relapse or death from any cause. The probability of RFS will be estimated using the Kaplan-Meier method. Median RFS (range) and 95% CI will be calculated
8. Progression-free survival, defined as the time elapsed since treatment initiation until disease progression or death from any cause. | 2010-2022
  PFS will be calculated as the time elapsed since treatment initiation until disease progression or death from any cause. Patients will be censored at the date of last follow-up if still alive or without disease progression at the time of the analysis. The probability of PFS will be estimated using the Kaplan-Meier method. Median PFS (range) and 95% CI will be calculated.
9. Percentage of patients with bleeding events an infections leading to hospitalization or death during the follow-up period. | 2010-2022
  A descriptive analysis will be performed on the bleeding episodes and/or infection reported during each treatment line received, including the absolute and relative frequencies and the corresponding 95% CI.

CONTACTS AND LOCATIONS:
Locations (1):
- Asociación Instituto Biodonostia, San Sebastián, Guipuzcoa, Spain

IPD SHARING:
Plan to Share IPD: Undecided